CLINICAL TRIAL: NCT00240045
Title: The Use of Midodrine, Octreotide and Albumin in Refractory Ascites
Brief Title: The Use of Drugs to Improve Kidney Function in Patients With Liver and Kidney Dysfunction
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Novartis (Industry)
Responsible Party: Dr. Vince Bain, University of Alberta
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VB-PG-007
Record Dates: First submitted 2005-10-13; First posted 2005-10-17 (Estimated); Last update posted 2007-12-06 (Estimated); Status verified 2005-10

CONDITIONS: Type 2 Hepatorenal Syndrome; Refractory Ascites
Keywords: Hepatorenal syndrome; Refractory ascites; Midodrine; Octreotide; Albumin; Cirrhosis
MeSH Terms: conditions — Ascites; Hepatorenal Syndrome; Fibrosis | interventions — Midodrine; Albumins; Octreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Midodrine, albumin, octreotide LAR; Drug: midodrine, octreotide, albumin

INTERVENTIONS:
Drug: Midodrine, albumin, octreotide LAR
Drug: midodrine, octreotide, albumin — midodrine up to 12.5 mg tid, octreotide LAR 20 mg im once, albumin 150 mg q weekly

SUMMARY:
We will address the hypothesis that refractory ascites and Type 2 hepatorenal syndrome are mediated in part by diminished circulatory volume and that treatment with midodrine, octreotide and albumin can improve renal and patient outcomes by restoring effective circulating volume and systemic perfusion.

Our primary objective is to assess change in creatinine clearance using inulin. We will enroll 15 patients with Type 2 hepatorenal syndrome or refractory ascites once inclusion and exclusion criteria are satisfied. They will be treated for 1 month with octreotide LAR, albumin and midodrine. Renal, serum and neurohormonal parameters will be measured before, during, and after initiation of drug and compared.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis (biopsy or compatible clinical (ascites, varices), laboratory (low albumin, elevated bilirubin, elevated INR) and radiologic data (nodular appearing liver on ultrasound)).

Type 2 hepatorenal syndrome and/or refractory ascites

Exclusion Criteria:

* Secondary causes of renal dysfunction (proteinuria >500 mg/day, active urinary sediment, abnormal renal ultrasound, nephrotoxic medications) Bacterial infection (positive blood, urine or ascites cultures) within the past 2 weeks Gastrointestinal hemorrhage or encephalopathy within the past 2 weeks Age <18 Transvenous intrahepatic portosystemic stent shunt (TIPS) Hepatocellular carcinoma beyond the Milan criteria

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2005-10; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Improvement in renal function (creatinine) | one month

SECONDARY OUTCOMES:
Ascites control | one month

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Bain, MD, FRCPC, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada